CLINICAL TRIAL: NCT04225377
Title: Observational Study of Physical Therapy Combined With Adapted Education on Physical Fitness in College Students With Physical Disabilities
Brief Title: Physical Therapy Combined With Adapted Education on Physical Fitness in College Students With Physical Disabilities
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: Yueh Ling Hsieh's laboratory funding (Unknown)
Responsible Party: Sponsor
Other Study IDs: CRREC-108-134
Record Dates: First submitted 2020-01-04; First posted 2020-01-13 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Physical Fitness Performance of Students With Physical and Mental Disabilities; Physical Therapy Technology Integrated Into Physical Education Curriculum
Keywords: adapted physical education,Physical Therapy,physical fitness,disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To integrate therapeutic exercise and techniques of physical therapy into adapted physical education courses to improve the limitations and obstacles of the physical body, and health-related physical fitness training and physical therapy into adapted physical education courses to improve the limitations and obstacles of the physical body and to improve the physical fitness performance of the students with physical and mental disabilities. Expected results: Adapting to physical education curriculum supplemented by physical therapy techniques can effectively improve the degree of physical and mental impairment, the effect of add-on fitness training, and make the physical fitness performance of students with physical and mental disabilities more progressive.

DETAILED DESCRIPTION:
Background: The degree of disorder of college students with physical and mental disabilities over 18 years old is mostly chronic, and the disease may be stable, the body and mind are more adaptable to their own disability, but also due to physical disorders, health-related physical fitness can enter the process of degradation earlier than the average person. Students with physical and mental disabilities can increase physical activity by adapted physical education courses, but because of their individual differences, the degree of disorder and the category are different. It is difficult to progress physical fitness without further professional intervention. Therefore, if the physiotherapy exercise therapy training and the hand-on treatment course are combined and integrated into the adapted physical education course and after-school time, it will be able to effectively improve the physical fitness performance of students with physical and mental disabilities. Purpose: To integrate therapeutic exercise and techniques of physical therapy into adapted physical education courses to improve the limitations and obstacles of the physical body, and health-related physical fitness training and physical therapy into adapted physical education courses to improve the limitations and obstacles of the physical body and to improve the physical fitness performance of the students with physical and mental disabilities. Methods: It is expected that 20-30 students and students over 18 years old who are involved in physical education classes will be recruited. One semester of physical education for a total of 18 weeks, 2 lessons per week (100 minutes), each class covers 40 minutes of individualized physical therapy sports therapy guidance and hand-on treatment and 40 minutes of group fitness training courses. The physical fitness assessment was conducted before the first week of each semester and after the 18th week. The "Physical Therapy and Adaptation to Physical Education" program was implemented for two semesters. The fitness assessment program mainly includes: cardio endurance, muscle fitness, body composition, softness and balance. Expected results: Adapting to physical education curriculum supplemented by physical therapy techniques can effectively improve the degree of physical and mental impairment, the effect of add-on fitness training, and make the physical fitness performance of students with physical and mental disabilities more progressive.

ELIGIBILITY:
Inclusion criteria

* College students whose body, mind and limbs are not suitable for strenuous exercise recognized by the Physical Education Office of China Medical University.
* College students with permanent or temporary physical and mental disabilities.
* College students with congenital disorders or temporary disorders.

Exclusion criteria

* Exercise will affect wound healing after surgery
* Medical order emphasize people who cannot exercise
* Certifiable disease
* Unable to follow the exercise command
* History of malignant tumors
* Any other factors that are unable to complete the exercise required in the course
* Subjects need to take matters in the Sports Safety Questionnaire project as a precaution

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 10 students of China Medical University will be recruited to take physical education courses (ages 18-25 years old), regardless of gender. Students who participate in the physical education courses are required to attach relevant certificates issued by the physician and sign the exercise safety consent form.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Posture assessment | 36weeks
  Using the plumb line to assess the subject's standing upright, whether the earlobe (mastoid process), acromion, middle torso, greater trochanter of femur, knee joint and lateral malleolus are on a vertical gravity line,whether the gravity line passes through the cervical, thoracic, lumbar and sacral vertebral concave posture assessment.

SECONDARY OUTCOMES:
Body composition | 36 weeks
  Body mass index(BMI)== kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
Muscle fitness/muscle endurance | 36 weeks
  The subject sits on a chair with the soles of both feet resting on the ground, holding dumbbells (8 pounds for men, 5 pounds for women) with arms straight and hanging down next to the chair. After the start, the subject will bend his arms to the shoulders and calculate 30 seconds. The total number of correct bends in a second.
  The subject sits in the middle of the chair with his back straight, hands crossed in front of his chest, after the start, the subject stands up and sits down, and counts the number of standing up and sitting times completed within 60 seconds.
Upper and lower limbs and body flexibility | 36 weeks
  The subject adopts a standing posture, with the dominant hand placed behind the shoulder on the same side, with the palm facing the back, with the fingers straight, stretch down as far as possible along the center of the back, and the palm of the other hand outwards from the bottom Extend your back upwards, keep your hands as close as possible, touch each other, or overlap your hands. Never hold and pull with your hands. Measure the distance between the middle finger of both hands.
  The subject sits on the front edge of the chair, with one foot bent on the ground, the other foot is straight forward, the heel touches the ground, the toes are raised, and the palms of both hands are folded (middle fingers) and stretched out. Stretch straight feet. Measure the distance from the middle finger to the toe.
  The subject is standing with both feet, the body bends forward, left and right, and then measures the distance from the middle finger to the ground.
Cardiopulmonary endurance | 36 weeks
  First measure the height of 1/2 of the line between the midpoint of the patella and the iliofemoral ridge of the subject, and mark it with colored tape on the wall or door frame as the basis for knee elevation. After the start, the subject should step on the spot as soon as possible, and the knee must be raised to the marked height. Record the number of steps completed in 2 minutes.
Agility | 36 weeks
  The chair needs to lean against the wall or rely on other safety objects. The subject sits on the chair, with both feet on the ground, one foot can be slightly forward, and the chair can be supported when getting up, but running is not allowed during the journey. The subject sits on a chair. After the start, the subject stands up and walks to the pyramid, walks around the pyramid and returns to the chair to sit down and calculate the required time.
Balance | 36 weeks
  Stand with your hands on your waist, stand on one foot, and place the foot off the ground on the inside of the ankle that supports your foot. Record the right and left foot support time for correct actions, with a full score of 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Ling Hsieh, PHD, Principal Investigator — China Medical University, China
Locations (2):
- Taiwan (2):
  - Department of Physical Therapy of China Medical University, Taichung, Test2
  - China Medical University, Taichung